CLINICAL TRIAL: NCT05779878
Title: Comparative Effects of Myofascial Arm Pull Technique and Post Isometric Relaxation on Pain, Range of Motion and Functional Disability in Adhesive Capsulitis After Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahreen Anwar (Other)
Responsible Party: Sponsor-Investigator, Sahreen Anwar, Dr, Riphah International University
Organization: Riphah International University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC_FSD_00319
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group A (Experimental): This group will be given Post isometric relaxation technique. Total intervention protocol will be given for four weeks of duration 3 sessions per week with total 12 sessions.
  Interventions: Other: Post Isometric Relaxation
- Interventional Group B (Experimental): This Group will be given myofascial arm pull technique . Total intervention protocol will be given for four weeks of duration 3 sessions per week with total 12 sessions.
  Interventions: Other: Myofascial arm pull technique

INTERVENTIONS:
Other: Post Isometric Relaxation — Post-isometric relaxation (PIR) is a soft tissue stretching technique used by many health care professionals to lengthen both acute and chronic short muscles.
  Arms: Interventional Group A
Other: Myofascial arm pull technique — Myofascial therapy is described as the promotion of psychophysiological, neurological and structural adaptive capability as multiplexed via the myofascial system. Fascia covers all body structures, particularly muscles and their constituent myofibrils
  Arms: Interventional Group B

SUMMARY:
Adhesive capsulitis (AC) also known as frozen shoulder typically manifests to decrease range of motion (ROM) and function and increase pain in shoulder .Objective of the study is To compare the effects of Myofascial Arm Pull Technique and Post-isometric Relaxation on Pain, Range of Motion and functional disability in adhesive capsulitis after mastectomy. The study design will be a Randomized Clinical Trial that will be used to compare the effects of Myofascial arm pull technique with post isometric relaxation. Subject with adhesive capsulitis meeting the predetermined inclusion & exclusion criteria will be divided into two groups. Pre assessment will be done using numeric pain rating scale NPRS for pain , shoulder pain and disability index (SPADI) tool for disability and Goniometer for Range of motion. Consent will be taken from patients by consent form the patients. They will be divided into two groups randomly by Random Number Generator table: Group A and Group B. For common treatment, both the groups will receive Ultrasound with a dosage of 1 MHz in frequency, continuous mode and 1.5 W/ cm2 of intensity for 10 minutes of treatment duration and Movement with mobilization will be applied for 15 times in 3 sets, and a 1- minute rest period was provided between each set. Group A will be given Post isometric relaxation technique with ultrasonic therapy. Group B will be given myofascial arm pull technique with ultrasonic. Total intervention protocol will be given for four weeks of duration 3 sessions per week with total 12 sessions. In Post isometric relaxation technique the therapist will slowly provide resistance in the direction of flexion, abduction, or external rotation, and without the subject intending to move for 15 minutes/ day, 3 times/week for 12 weeks. Similarly, myofascial arm pull technique the therapist will hold arm of the subject firmly and initial stretch will be applied in abduction and external rotation for 8-10 times in each session per day for 3 days/week for 4 weeks. Outcome measures will be measured at baseline, after 2 weeks and after 4 weeks. Data analysis will be done by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Only Female gender
* Age between 25 to 50 years with post mastectomy.
* Diagnosis of breast cancer (grade 1to3 b).
* Post mastectomy state at least 6 months.
* Shoulder pain that began after the breast cancer surgery

Exclusion Criteria:

* Bilateral breast cancer.
* History of neurologic deficits affecting shoulder functioning during daily activites.
* On numeric pain rating scale pain will be less than 5.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-06-09 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain in Shoulder Joint | 4 weeks
  Pain will be measured by using Numeric pain rating scale
Range of motion in all planes | 4 weeks
  Range of motions in all planes will be measured by using goniometer
Functional disability | 4 weeks
  Functional disability will be measured by using Shoulder Pain and Disability Index

CONTACTS AND LOCATIONS:
Locations (1):
- Allied Hospital, Faisalābad, Punjab Province, Pakistan